CLINICAL TRIAL: NCT00377052
Title: A Phase II Study of Bortezomib and Gemcitabine in Patients With Relapsed Mantle Cell Lymphoma
Brief Title: Bortezomib and Gemcitabine in Treating Patients With Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I172; CAN-NCIC-IND172 (Registry Identifier: PDQ); ORTHO-CAN-NCIC-IND172 (Other: Ortho Biotech); CDR0000493021 (Other: PDQ); B9E-CA-0485 (Other: Lilly)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma
Keywords: recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Bortezomib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bortezomib + Gemcitabine (Experimental)
  Interventions: Drug: bortezomib; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bortezomib — 1.0 mg/m2 IV; injection bolus (3-5 sec) Twice weekly x 2 weeks every three weeks
Drug: gemcitabine hydrochloride — 1000 mg/m2 IV; injection 30 minute infusion Once weekly x 2 weeks every three weeks

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may help gemcitabine work better by making cancer cells more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving bortezomib together with gemcitabine works in treating patients with relapsed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy (response rate) of bortezomib and gemcitabine hydrochloride in patients with relapsed mantle cell lymphoma.
* Determine the toxicity of this regimen in these patients.
* Determine the time to progression and duration of response in patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive bortezomib IV on days 1, 4, 8, and 11 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter until relapse/progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma

  * Relapsed disease
* Not refractory to prior therapy

  * Must have received 1-3 prior systemic chemotherapy regimens AND has had no disease progression while receiving chemotherapy or within 1 month of last dose of most recent therapy
* Clinically and/or radiologically documented disease

  * At least 1 site of disease must be bidimensionally measurable by CT scan or MRI with ≥ 1 lesion meeting 1 of the following criteria:

    * Lymph nodes ≥ 1.5 cm x 1.5 cm by spiral CT scan
    * Non-nodal lesion ≥ 1 cm x 1 cm by MRI, CT scan, or physical exam
  * No nonmeasurable disease only
* No preexisting ascites or pleural effusion ≥ grade 2
* No known CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST or ALT ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF ≥ 45% by echocardiogram or MUGA
* No history of allergic reactions attributed to compounds containing boron or mannitol
* No preexisting edema ≥ grade 2
* No preexisting neuropathy (sensory and/or pain) ≥ grade 2
* No preexisting shortness of breath ≥ grade 2
* No history of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No other serious illness or medical condition that would preclude compliance with study requirements, including any of the following:

  * Serious uncontrolled infection
  * Uncontrolled or severe cardiovascular disease, including any of the following:

    * Myocardial infarction within the past 6 months
    * New York Heart Association class III-IV heart failure
    * Uncontrolled angina
    * Clinically significant pericardial disease
    * Cardiac amyloidosis
  * Significant neurological disorder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior chemotherapy
* No prior radioactive monoclonal antibody therapy
* No prior bortezomib
* No prior investigational therapy (except for flavopiridol)
* No prior radiotherapy to > 25% of functioning bone marrow
* At least 4 weeks since prior radiotherapy and recovered

  * Low-dose, nonmyelosuppressive radiotherapy may be allowed
* At least 2 weeks since prior major surgery
* No other concurrent anticancer therapy
* No concurrent corticosteroids
* No other concurrent cytotoxic chemotherapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-01-16 (Actual); Primary Completion 2009-04-21 (Actual); Study Completion 2011-06-21 (Actual)

PRIMARY OUTCOMES:
Objective tumor response (overall response rate with 95% confidence interval) | each cycle
Time to progression at median time | each cycle and every 3 months after treatment
Duration of response (median and range) | each cycle and every 3 months after treatment
Rate of stable disease and progressive disease | each cycle and every 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: C. Tom Kouroukis, MD, Principal Investigator — Margaret and Charles Juravinski Cancer Centre
Locations (11):
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - QEII, CCR, Hematology Research, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University - Dept. Oncology, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kouroukis CT, Fernandez LA, Crump M, Gascoyne RD, Chua NS, Buckstein R, Turner R, Assouline S, Klasa RJ, Walsh W, Powers J, Eisenhauer E. A phase II study of bortezomib and gemcitabine in relapsed mantle cell lymphoma from the National Cancer Institute of Canada Clinical Trials Group (IND 172). Leuk Lymphoma. 2011 Mar;52(3):394-9. doi: 10.3109/10428194.2010.546015. PMID 21323520